CLINICAL TRIAL: NCT00831194
Title: Stress, Dietary Lapse and Weight Loss Among Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lawrence J. Cheskin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB#00001685
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Type 2 Diabetes; Obesity; Weight loss; PDA; Stress; Dietary lapse; salivary alpha amylase
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet plan and PDA (Experimental)
  Interventions: Behavioral: Personalized diet plan and PDA self reporting.

INTERVENTIONS:
Behavioral: Personalized diet plan and PDA self reporting. — Participants will be given personalized diet plan with a 0.5- 1 lb weight loss/week, based on each person's goals. He/she will also be prompted by a pre programmed PDA to enter dietary lapses and stress inducing events. Saliva samples will be collected as per the study plan.

SUMMARY:
A clinical trial that uses personal digital assistants (PDAs) to assist in examining the relationship between self reported stress, an objective biochemical indicator of stress (salivary alpha amylase) and self-reported dietary lapse among type 2 diabetic adults who are interested/undergoing in weight loss.

DETAILED DESCRIPTION:
In the study, all participants will be provided with a personalized ADA-based diet plan and a pre-programmed PDA. They will be required to record their mood and activities into the PDA whenever PDA prompts, they break their diet plan, and/or and face significant stress. They will also be required to collect saliva samples periodically. In addition to this they will be administered the Trier Social Stress Test once during the study, where they will perform certain stress inducing tasks like delivering a speech and solving maths problems. Salivary samples will be collected before and after these tasks. They will also take various questionnaires during each of the 15 to 16 visits. The completed questionnaires, PDA records and reports of salivary alpha amylase levels will be analyzed to examine the corelation between stress, dietary lapse and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 65 years, seeking weight loss.
* Type 2 diabetes diagnosis by American Diabetes Association standard criteria. (Confirmed by physician's note or blood glucose reports in previous year or Prescriptions for medications to control blood glucose dated in participant's name within last year).
* BMI > 30 kg/m2.

Exclusion Criteria:

* Major depression.
* Cognitive impairment severe enough to preclude informed consent or valid self report.
* Use of medications that significantly affect appetite.
* Eating disorder.
* Inability or unwillingness to use PDA for 6 months.
* Inability or unwillingness to collect saliva samples.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Self reported stress, weight loss, and salivary alpha amylase. | 1 year

SECONDARY OUTCOMES:
Positive correlation between levels of salivary alpha amylase (sAA) and weight loss, BMI and levels of sAA, levels of sAA and maladaptive coping. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States